CLINICAL TRIAL: NCT06724744
Title: Effect of Manual Diaphragmatic Release on Ventilatory Functions and Functional Capacity in Elderly Diabetic Women
Brief Title: Manual Diaphragmatic Release on Ventilatory Functions in Elderly Diabetic Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Saad, Assistant Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Manual Diaphragmatic Release
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Diabetes; Elderly
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual diaphragmatic release group (Active Comparator): 30 elderly diabetic women participating in manual diaphragmatic release plus aerobic training
  Interventions: Other: Aerobic training; Other: Manual Diaphragm Release
- Control group (Active Comparator): 30 elderly diabetic women participating in aerobic training only
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: Aerobic training — For twelve weeks, the women participate in aerobic training on cycle ergometer. Each session consists of 30-45 minutes of cycling at a moderate intensity, accompanied by a workout heart rate ranging from 65% to 75% of the maximal heart rate and ranging between 12 and 14 on the Borg rating of perceived exertion 20-point scale. After ten minutes of warm-up, every session ends with a brief 3-minute period of cool-down.
Other: Manual Diaphragm Release — The participant is asked assume a supine position with relaxed limbs. The therapist should position themselves at the head of the participant and make manual contact with the pisiform, hypothenar region, and the last three fingers on both sides, underneath the seventh to tenth rib costal cartilages. The therapist's forearms should be aligned towards the participant's shoulders. During the inspiratory phase, the therapist gently pulled the points of contact with both hands in the direction of the head and slightly laterally, accompanying the elevation of the ribs. Therapist progressively increases the depth of their contact within the costal margin.
  Arms: Manual diaphragmatic release group

SUMMARY:
Evaluate the effect of manual diaphragmatic release on ventilatory functions and functional capacity in elderly diabetic women.

DETAILED DESCRIPTION:
Sixty elderly type 2 diabetic women were sourced from the endocrinology outpatient clinic at Mansoura University hospitals in Egypt, with referrals from endocrinologists. Patients were randomly assigned into two groups.

The study group includes 30 women participating in manual diaphragmatic release plus aerobic training for 12 weeks, while the control group includes 30 women participating in aerobic training only for 12 weeks. At baseline and poststudy, the following outcomes are assessed:

1. Ventilatory functions (Forced vital capacity and forced expiratory volume in the first second).
2. Functional capacity using modified Bruce treadmill incremental exercise test (Maximal oxygen consumption estimation).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic for more than 5 years.
* Well controlled diabetes with glycated hemoglobin≤7%.
* Normal to mild ventilatory functions impairment.
* Their ages ranges from 65 to 70 years old.
* Their body mass index are less than 30 Kg/m2.

Exclusion Criteria:

* Other types of diabetes.
* Patients with any other chronic chest diseases .
* Cardiovascular disorders (coronary heart disease, heart failure, cardiac arrhythmia, peripheral arterial disease, uncontrolled hypertension).
* Smokers.
* Rheumatoid arthritis.
* Musculoskeletal/ neurological limitations to exercise.

Ages: 65 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Females
Enrollment: 60 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Ventilatory functions | At baseline and after 12 weeks
  Ventilatory function parameters, including forced vital capacity and forced expiratory volume in the first second are measured by experienced technicians at baseline and after 12 weeks in all groups using the Medgraphics pulmonary function testing system (Breezesuite Ultima PFX, Milano, Italy) in strict adherence to the guidelines outlined in the user manual.

SECONDARY OUTCOMES:
Functional capacity | At baseline and after 12 weeks
  Cardiopulmonary exercise test will be conducted for all women at baseline and post-study based on the guidelines set by the American College of Sports Medicine to determine maximal oxygen consumption for each women.

CONTACTS AND LOCATIONS:
Overall Officials: Saher Lotfy Elgayar, Ph.D, Study Director — Department of Physiotherapy Faculty of Allied Medical Sciences Middle East University Amman Jordan
Locations (1):
- Endocrinology outpatient clinic at Mansoura University, Al Mansurah, Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: No